CLINICAL TRIAL: NCT05204420
Title: Spontaneous Gastric Intramural Hematoma: Case Report and Literature Review
Status: Completed | Type: Observational
Sponsor: University of Balamand (Other)
Responsible Party: Principal Investigator, Omar Tabbikha, General Surgery Resident, University of Balamand
Other Study IDs: UBalamand
Record Dates: First submitted 2022-01-12; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Gastric Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Gastric wide local excision for bleeding mass — Laparoscopic partial gastrectomy for gastric submucosal mass

SUMMARY:
Patient previously healthy found to have spontaneous gastric intramural hematoma

DETAILED DESCRIPTION:
28 year old male patient previously healthy presented with diarrhea and diffuse abdominal pain of 1 week duration that exacerbated 1 day prior to presentation. CT showed anterior abdominal mass possibly from the outer gastric wall. Gastroscopy suspected a submucosal tumor in the body and antrum. Patient's pain exacerbated and developed drop in hemoglobin. Urgent CT scan showed a bleeding gastric tumor. Urgent laparotomy identified a bleeding gastric lesion at greater curvature. Partial gastrectomy done with abutting mesocolon resection. Surgical specimen pathology showed gastric intramural hematoma that was considered spontaneous.

ELIGIBILITY:
Inclusion Criteria:

* any patient presenting with gastric bleeding tumors

Exclusion Criteria:

* patients on anticoagulants and patient with gastric medical history

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously healthy presenting with bleeding gastric mass
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Spontaneous gastric intramural hematoma | 1 month
  Spontaneous gastric intramural hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Omar Tabbikha, MD, Principal Investigator — University of Balamand
Locations (1):
- University of Balamand, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
Publishing a case report of our finding